CLINICAL TRIAL: NCT01667679
Title: A Randomized, Double-Blind, Double-Dummy, Active-Controlled, Cross-Over Study Evaluating the Efficacy and Safety of 20 mg Sumatriptan Powder Delivered Intranasally With the Bi-directional Device Compared With 100 mg Sumatriptan Tablets in Adults With Acute Migraine With or Without Aura
Brief Title: Efficacy and Safety of 20 mg Sumatriptan Powder Delivered Intranasally With the Bi-directional Device Compared With 100 mg Sumatriptan Tablets in Adults With Acute Migraine With or Without Aura
Acronym: COMPASS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Avanir Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: OPN-SUM-MIG-3302
Record Dates: First submitted 2012-08-06; First posted 2012-08-17 (Estimated); Results first posted 2017-03-14 (Actual); Last update posted 2017-04-12 (Actual); Status verified 2017-03

CONDITIONS: Migraine; Headaches
Keywords: Migraine; Headaches; Sumatriptan
MeSH Terms: conditions — Migraine Disorders; Headache | interventions — Sumatriptan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- OPTINOSE SUMATRIPTAN and Placebo (Experimental): 20 mg OPTINOSE SUMATRIPTAN Powder Delivered Intranasally With the Bi-directional Device nasally and Placebo Tablet
  Interventions: Drug: OPTINOSE SUMATRIPTAN delivered nasally and placebo tablet
- 100mg Sumatriptan and OPTINOSE Placebo (Active Comparator): 100 mg Sumatriptan Tablet and OPTINOSE Placebo delivered nasally
  Interventions: Drug: 100 mg Sumatriptan Tablet and OPTINOSE Placebo delivered nasally

INTERVENTIONS:
Drug: 100 mg Sumatriptan Tablet and OPTINOSE Placebo delivered nasally
  Arms: 100mg Sumatriptan and OPTINOSE Placebo
Drug: OPTINOSE SUMATRIPTAN delivered nasally and placebo tablet
  Arms: OPTINOSE SUMATRIPTAN and Placebo

SUMMARY:
This study is being conducted to determine if OPTINOSE SUMATRIPTAN delivered nasally (through the nose) using the OPTINOSE SUMATRIPTAN DEVICE can reduce the pain associated with migraine headaches in 30 minutes after use.

DETAILED DESCRIPTION:
The primary objective for this study is to compare the proportion of attacks in which pain reduction (defined as a decrease in pain intensity of at least 1 point) is achieved at 30 minutes following 20 mg OPTINOSE SUMATRIPTAN treatment with 100 mg Sumatriptan Tablets

ELIGIBILITY:
Inclusion Criteria:

* Man or woman, between the ages of 18 to 65 years, inclusive at screening
* Have a diagnosis of episodic migraine, with or without aura according to InternationalClassification of Headache Disorders (2nd Edition) (ICHD-2) for at least 1 year prior to screening
* Experiences between 2 and 8 migraine attacks per month for the past 12 months
* Women of child bearing potential must be practicing an effective method of birth control
* Women of child-bearing potential must have a negative urine pregnancy test at the screening visit and a negative urine pregnancy test at the randomization visit
* Demonstrate the ability to use the bi-directional delivery device correctly
* Able and willing to read and comprehend written instructions and complete the electronic diary information required by the protocol
* Must be capable, in the opinion of the Investigator, of providing informed consent to participate in the study. Subjects (and their legally acceptable representatives, if applicable) must sign an informed consent document indicating that they understand the purpose of and procedures required for the study and are willing to participate in the study

Exclusion Criteria:

* Inability to distinguish other headaches from migraine
* Experiences headache of any kind at a frequency greater than or equal to 15 days per month
* History of resistance to sumatriptan, or non-response to 2 or more other triptans, defined as subjects who have not responded to an adequate dose and duration of treatment
* Current use of medication for migraine prophylaxis that has not been stable (no dose adjustment) for 30 days prior to screening
* Chronic opioid therapy (>3 consecutive days in the 30 days prior to screening)
* Current treatment with monoamine oxidase A (MAO-A) inhibitors or use within 4 weeks before randomization
* Have hemiplegic or basilar migraine
* History, symptoms or signs of ischemic cardiac, cerebrovascular or peripheral vascular syndromes. Ischemic cardiac syndromes include, but are not limited to, angina pectoris of any type (e.g., stable angina of effort, vasospastic forms of angina such as the Prinzmetal variant), all forms of myocardial infarction and silent myocardial ischemia. Cerebrovascular syndromes include, but are not limited to, strokes of any type as well as transient ischemic attacks. Peripheral vascular disease includes, but is not limited to, ischemic bowel disease, Raynaud syndrome
* Uncontrolled hypertension (screening systolic/diastolic blood pressure >140/95 mmHg)
* Have severe hepatic impairment
* Have history of epilepsy or conditions associated with a lowered seizure threshold
* History (within 2 years) of drug or alcohol abuse as defined by Diagnostic and Statistical Manual of Mental Disorders 4th edition (DSM-IV) criteria

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 275 (Actual)
Dates: Start 2012-08; Primary Completion 2014-03 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (13):
- United States (13):
  - San Francisco Clinical Research Center, San Francisco, California
  - California Medical Clinic for Headache, Santa Monica, California
  - Associated Neurologists of Southern CT, P.C., Fairfied, Connecticut
  - Premiere Research Institute, West Palm Beach, Florida
  - MedVadis, Watertown, Massachusetts
  - Michigan Head and Pain Institute, Ann Arbor, Michigan
  - ClinVest, Springfield, Missouri
  - Mercy Health Research, St Louis, Missouri
  - DENT Neurologic Institute, Amherst, New York
  - Headache Welness Center, Greensboro, North Carolina
  - PMG Research of Winston Salem, LLC, Winston-Salem, North Carolina
  - Jefferson Headache Center, Philadelphia, Pennsylvania
  - Coastal Carolina Research Center, Mt. Pleasant, South Carolina

REFERENCES:
- [Derived] Lipton RB, McGinley JS, Shulman KJ, Wirth RJ, Buse DC. Faster Improvement in Migraine Pain Intensity and Migraine-Related Disability at Early Time Points with AVP-825 (Sumatriptan Nasal Powder Delivery System) versus Oral Sumatriptan: A Comparative Randomized Clinical Trial Across Multiple Attacks from the COMPASS Study. Headache. 2017 Nov;57(10):1570-1582. doi: 10.1111/head.13165. Epub 2017 Sep 7. PMID 28880380
- [Derived] Tepper SJ, Cady RK, Silberstein S, Messina J, Mahmoud RA, Djupesland PG, Shin P, Siffert J. AVP-825 breath-powered intranasal delivery system containing 22 mg sumatriptan powder vs 100 mg oral sumatriptan in the acute treatment of migraines (The COMPASS study): a comparative randomized clinical trial across multiple attacks. Headache. 2015 May;55(5):621-35. doi: 10.1111/head.12583. Epub 2015 May 4. PMID 25941016

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 334 participants were assessed for eligibility; of these, 275 participants were randomized.
Groups:
- 20 mg Sumatriptan+PBO (TP1)/100 mg Sumatriptan+PBO (TP2): In Treatment Period (TP) 1 (<=12 weeks), participants received 20 milligrams (mg) sumatriptan nasal powder delivered intranasally with a bi-directional device and a placebo (PBO) tablet taken orally. After completing Treatment Period 1 (upon reaching 12 weeks or treating the fifth qualifying migraine headache in the treatment period, whichever came first), participants entered Treatment Period 2 (<=12 weeks), during which they received a 100 mg sumatriptan tablet taken orally and placebo (lactose) as a nasal powder administered into the nostril on the side of the migraine, followed by another administration into the other nostril. Participants were to treat <=5 qualifying migraine headaches during Treatment Period 2.
- 100 mg Sumatriptan+PBO (TP1)/20 mg Sumatriptan+PBO (TP2): In Treatment Period 1 (<=12 weeks), participants received a 100 mg sumatriptan tablet taken orally and placebo (lactose) as a nasal powder administered into the nostril on the side of the migraine, followed by another administration into the other nostril. After completing Treatment Period 1 (upon reaching 12 weeks or treating the fifth qualifying migraine headache in the treatment period, whichever came first), participants entered Treatment Period 2 (<=12 weeks), during which they received 20 mg sumatriptan nasal powder delivered intranasally with a bi-directional device and a placebo tablet taken orally. Participants were to treat <=5 qualifying migraine headaches during Treatment Period 2.
Period: Treatment Period 1 (<=12 Weeks)
Arm/Group | 20 mg Sumatriptan+PBO (TP1)/100 mg Sumatriptan+PBO (TP2) | 100 mg Sumatriptan+PBO (TP1)/20 mg Sumatriptan+PBO (TP2)
Started | 138 | 137
Completed | 122 | 107
Not Completed | 16 | 30
Not completed — Failure to Treat Migraine Headache | 2 | 6
Not completed — Dosed Incorrectly | 2 | 0
Not completed — Lack of Efficacy | 2 | 0
Not completed — Could Not Tolerate Diary | 1 | 0
Not completed — Withdrawal by Subject | 6 | 13
Not completed — Adverse Event | 3 | 3
Not completed — Lost to Follow-up | 0 | 2
Not completed — Protocol Violation | 0 | 2
Not completed — Non-compliance | 0 | 3
Not completed — Moved Out of State | 0 | 1
Period: Treatment Period 2 (<=12 Weeks)
Arm/Group | 20 mg Sumatriptan+PBO (TP1)/100 mg Sumatriptan+PBO (TP2) | 100 mg Sumatriptan+PBO (TP1)/20 mg Sumatriptan+PBO (TP2)
Started | 122 | 107
Completed | 100 | 85
Not Completed | 22 | 22
Not completed — Withdrawal by Subject | 6 | 4
Not completed — Non-compliance with Electronic Diary | 2 | 0
Not completed — Lost to Follow-up | 8 | 10
Not completed — Non-compliance | 3 | 4
Not completed — Sponsor Decision | 1 | 0
Not completed — Failure to Treat Migraine Headache | 1 | 0
Not completed — Adverse Event | 1 | 0
Not completed — Significant Improvement in Migraine | 0 | 1
Not completed — Partially Dosed | 0 | 1
Not completed — Brought in before 12 Weeks/5 Migraines | 0 | 1
Not completed — Refused Last Day of Visit 4 Procedures | 0 | 1

BASELINE CHARACTERISTICS:
Population: Baseline data are reported for participants in the Safety Analysis Set, defined as all randomized participants who received at least one dose of sumatriptan (20 mg nasal powder or 100 mg tablet).
Groups:
- 20 mg Sumatriptan+PBO (TP1)/100 mg Sumatriptan+PBO (TP2): In Treatment Period 1 (<=12 weeks), participants received 20 milligrams (mg) sumatriptan nasal powder delivered intranasally with a bi-directional device and a placebo (PBO) tablet taken orally. After completing Treatment Period 1, participants entered Treatment Period 2 (<=12 weeks), during which they received a 100 mg sumatriptan tablet taken orally and placebo (lactose) as a nasal powder administered into the nostril on the side of the migraine, followed by another administration into the other nostril.
- 100 mg Sumatriptan+PBO (TP1)/20 mg Sumatriptan+PBO (TP2): In Treatment Period 1 (<=12 weeks), participants received a 100 mg sumatriptan tablet taken orally and placebo (lactose) as a nasal powder administered into the nostril on the side of the migraine, followed by another administration into the other nostril. After completing Treatment Period 1, participants entered Treatment Period 2 (<=12 weeks), during which they received 20 mg sumatriptan nasal powder delivered intranasally with a bi-directional device and a placebo tablet taken orally.
- Total: Total of all reporting groups
Arm/Group | 20 mg Sumatriptan+PBO (TP1)/100 mg Sumatriptan+PBO (TP2) | 100 mg Sumatriptan+PBO (TP1)/20 mg Sumatriptan+PBO (TP2) | Total
Number analyzed (Participants) | 133 | 129 | 262
Age, Continuous [Mean (Standard Deviation); unit: Years] | 39.5 (12.55) | 40.7 (11.93) | 40.1 (12.24)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 107 | 115 | 222
  Male | 26 | 14 | 40
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 3 | 1 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 24 | 26 | 50
  White | 104 | 100 | 204
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 2 | 4

OUTCOME MEASURES:

1. Primary Outcome: Mean Sum of Migraine Pain Intensity Differences (SPID)-30
Description: SPID-30 is defined as the sum of the pain intensity differences (measured as area under the curve) from dosing (Baseline) through 30 minutes post-dose for headaches with a Baseline intensity of mild, moderate, or severe. The range of possible scores is -60 to +90. A higher number indicates a greater reduction in pain intensity. Negative values indicate worsening pain. A value of "0" indicates that there was no change in pain intensity from Baseline through 30 minutes. Results are from an analysis of covariance (ANCOVA) model with treatment, period, and treatment sequence as fixed effects and participant as a random effect. The Last Observation Carried Forward (LOCF) imputation method (missing values were replaced by carrying forward the preceding value) was used for this analysis.
Time Frame: Baseline and 30 minutes post-dose (up to 24 weeks)
Population: Full Analysis Set (FAS): all participants who experienced at least 1 headache attack per treatment period, received at least 1 dose of study medication (sumatriptan nasal powder or tablet) in each treatment period, and had at least 1 post-Baseline assessment for a treated attack in each treatment period.
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Groups:
- 20 mg Sumatriptan Nasal Powder: Participants received 20 mg sumatriptan nasal powder delivered intranasally with a bi-directional device in Treatment Period 1 or Treatment Period 2.
- 100 mg Sumatriptan Tablet: Participants received a 100 mg sumatriptan tablet taken orally in Treatment Period 1 or Treatment Period 2.
Arm/Group | 20 mg Sumatriptan Nasal Powder | 100 mg Sumatriptan Tablet
Number analyzed (Participants) | 185 | 185
scores on a scale | 10.80 (0.880) | 7.41 (0.880)
Statistical Analysis 1: Comparison: 20 mg Sumatriptan Nasal Powder vs 100 mg Sumatriptan Tablet; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = 3.39, 95% CI 2-sided [1.76 to 5.01], Standard Error of Mean 0.824

2. Secondary Outcome: Mean Sum of Migraine Pain Intensity Differences (SPID)-30 for Headaches With a Baseline Intensity of Mild and Moderate/Severe
Description: SPID-30 is defined as the sum of the pain intensity differences (measured as area under the curve) from dosing (Baseline) through 30 minutes post-dose for headaches with a Baseline intensity of mild and moderate/severe (rated on a 4-point scale: 0=none, 1=mild, 2=moderate, and 3=severe). The range of possible scores for all participants is -60 to +90. For participants with a mild headache at Baseline, the SPID range is -60 to +30. For participants with a moderate/severe headache at Baseline, the SPID range is -30 to +90. A higher number indicates a greater reduction in pain intensity. Negative values indicate worsening pain. A value of "0" indicates that there was no change in pain intensity from Baseline through 30 minutes. Results are from an ANCOVA model with treatment, period, and treatment sequence as fixed effects and participant as a random effect. The LOCF imputation method (missing values were replaced by carrying forward the preceding value) was used for this analysis.
Time Frame: Baseline and 30 minutes post-dose (up to 24 weeks)
Population: FAS. Only those participants with the type of attack specified were analyzed (specified by n=X, X in the corresponding category title). A single participant could have had both a mild and a moderate/severe attack.
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | 20 mg Sumatriptan Nasal Powder | 100 mg Sumatriptan Tablet
Number analyzed (Participants) | 185 | 185
scores on a scale
  mild attacks, n=113, 109 | 3.90 (0.921) | 0.24 (0.931)
  moderate/severe attacks, n=158, 168 | 13.83 (1.022) | 10.07 (0.997)
Statistical Analysis 1: Comparison: 20 mg Sumatriptan Nasal Powder vs 100 mg Sumatriptan Tablet; Test type: Superiority or Other; p = 0.0013, ANCOVA; Mean Difference (Final Values) = 3.66, 95% CI 2-sided [1.47 to 5.85], Standard Error of Mean 1.105 — mild attacks
Statistical Analysis 2: Comparison: 20 mg Sumatriptan Nasal Powder vs 100 mg Sumatriptan Tablet; Test type: Superiority or Other; p = 0.0002, ANCOVA; Mean Difference (Final Values) = 3.76, 95% CI 2-sided [1.84 to 5.68], Standard Error of Mean 0.971 — moderate/severe attacks

3. Secondary Outcome: Percentage of Attacks in Which Pain Reduction Was Achieved
Description: Percentage of attacks in which pain reduction (defined as a decrease in pain intensity of at least one point on the following scale: 0, none; 1, mild; 2, moderate; 3, severe) was achieved at 10, 15, 30, 45, 60, 90, and 120 minutes after the initial dose for all attacks.
Time Frame: 10, 15, 30, 45, 60, 90, and 120 minutes
Population: FAS. The LOCF imputation method was used in this analysis.
Measure: Number; unit: percentage of attacks
Units Other Than Participants: number of attacks
Arm/Group | 20 mg Sumatriptan Nasal Powder | 100 mg Sumatriptan Tablet
Number analyzed (Participants) | 185 | 185
Number analyzed (number of attacks) | 765 | 766
percentage of attacks
  10 minutes post-dose | 11.5 | 10.2
  15 minutes post-dose | 26.4 | 19.6
  30 minutes post-dose | 49.0 | 35.2
  45 minutes post-dose | 60.7 | 49.9
  60 minutes post-dose | 67.2 | 59.8
  90 minutes post-dose | 74.6 | 69.8
  120 minutes post-dose | 78.0 | 75.2
Statistical Analysis 1: Comparison: 20 mg Sumatriptan Nasal Powder vs 100 mg Sumatriptan Tablet; Test type: Superiority or Other; p = 0.3549, ANCOVA; Odds Ratio (OR) = 1.16, 95% CI 2-sided [0.85 to 1.60] — 10 minutes post-dose
Statistical Analysis 2: Comparison: 20 mg Sumatriptan Nasal Powder vs 100 mg Sumatriptan Tablet; Test type: Superiority or Other; p = 0.0005, ANCOVA; Odds Ratio (OR) = 1.51, 95% CI 2-sided [1.20 to 1.90] — 15 minutes post-dose
Statistical Analysis 3: Comparison: 20 mg Sumatriptan Nasal Powder vs 100 mg Sumatriptan Tablet; Test type: Superiority or Other; p < 0.0001, ANCOVA; Odds Ratio (OR) = 1.79, 95% CI 2-sided [1.45 to 2.21] — 30 minutes post-dose
Statistical Analysis 4: Comparison: 20 mg Sumatriptan Nasal Powder vs 100 mg Sumatriptan Tablet; Test type: Superiority or Other; p = 0.0002, ANCOVA; Odds Ratio (OR) = 1.56, 95% CI 2-sided [1.24 to 1.96] — 45 minutes post-dose
Statistical Analysis 5: Comparison: 20 mg Sumatriptan Nasal Powder vs 100 mg Sumatriptan Tablet; Test type: Superiority or Other; p = 0.0057, ANCOVA; Odds Ratio (OR) = 1.37, 95% CI 2-sided [1.10 to 1.71] — 60 minutes post-dose
Statistical Analysis 6: Comparison: 20 mg Sumatriptan Nasal Powder vs 100 mg Sumatriptan Tablet; Test type: Superiority or Other; p = 0.0654, ANCOVA; Odds Ratio (OR) = 1.26, 95% CI 2-sided [0.99 to 1.61] — 90 minutes post-dose
Statistical Analysis 7: Comparison: 20 mg Sumatriptan Nasal Powder vs 100 mg Sumatriptan Tablet; Test type: Superiority or Other; p = 0.2894, ANCOVA; Odds Ratio (OR) = 1.15, 95% CI 2-sided [0.89 to 1.49] — 120 minutes post-dose

4. Secondary Outcome: Percentage of Attacks in Which Pain Freedom Was Achieved
Description: Percentage of attacks in which pain freedom (defined as pain level reduced to none [Grade 0]) was achieved at 10, 15, 30, 45, 60, 90, and 120 minutes after the initial dose for all attacks.
Time Frame: Baseline and 10, 15, 30, 45, 60, 90, and 120 minutes post-dose (up to 24 weeks)
Population: FAS. The LOCF imputation method was used for this analysis.
Measure: Number; unit: percentage of attacks
Units Other Than Participants: number of attacks
Arm/Group | 20 mg Sumatriptan Nasal Powder | 100 mg Sumatriptan Tablet
Number analyzed (Participants) | 185 | 185
Number analyzed (number of attacks) | 765 | 766
percentage of attacks
  10 minutes post-dose | 2.5 | 1.3
  15 minutes post-dose | 7.2 | 3.7
  30 minutes post-dose | 18.2 | 10.8
  45 minutes post-dose | 31.0 | 21.3
  60 minutes post-dose | 41.2 | 32.9
  90 minutes post-dose | 52.8 | 44.9
  120 minutes post-dose | 60.4 | 56.3
Statistical Analysis 1: Comparison: 20 mg Sumatriptan Nasal Powder vs 100 mg Sumatriptan Tablet; Test type: Superiority or Other; p = 0.1771, ANCOVA; Odds Ratio (OR) = 1.85, 95% CI 2-sided [0.76 to 4.54] — 10 minutes post-dose
Statistical Analysis 2: Comparison: 20 mg Sumatriptan Nasal Powder vs 100 mg Sumatriptan Tablet; Test type: Superiority or Other; p = 0.0077, ANCOVA; Odds Ratio (OR) = 2.03, 95% CI 2-sided [1.21 to 3.42] — 15 minutes post-dose
Statistical Analysis 3: Comparison: 20 mg Sumatriptan Nasal Powder vs 100 mg Sumatriptan Tablet; Test type: Superiority or Other; p = 0.0003, ANCOVA; Odds Ratio (OR) = 1.82, 95% CI 2-sided [1.32 to 2.50] — 30 minutes post-dose
Statistical Analysis 4: Comparison: 20 mg Sumatriptan Nasal Powder vs 100 mg Sumatriptan Tablet; Test type: Superiority or Other; p < 0.0001, ANCOVA; Odds Ratio (OR) = 1.64, 95% CI 2-sided [1.29 to 2.09] — 45 minutes post-dose
Statistical Analysis 5: Comparison: 20 mg Sumatriptan Nasal Powder vs 100 mg Sumatriptan Tablet; Test type: Superiority or Other; p = 0.0016, ANCOVA; Odds Ratio (OR) = 1.41, 95% CI 2-sided [1.14 to 1.74] — 60 minutes post-dose
Statistical Analysis 6: Comparison: 20 mg Sumatriptan Nasal Powder vs 100 mg Sumatriptan Tablet; Test type: Superiority or Other; p = 0.0059, ANCOVA; Odds Ratio (OR) = 1.36, 95% CI 2-sided [1.09 to 1.69] — 90 minutes post-dose
Statistical Analysis 7: Comparison: 20 mg Sumatriptan Nasal Powder vs 100 mg Sumatriptan Tablet; Test type: Superiority or Other; p = 0.2717, ANCOVA; Odds Ratio (OR) = 1.14, 95% CI 2-sided [0.91 to 1.42] — 120 minutes post-dose

5. Secondary Outcome: Percentage of Attacks in Which Pain Relief Was Achieved
Description: Percentage of attacks treated at a severity of moderate (Grade 2) or severe (Grade 3) in which pain relief (defined as pain level reduced to none [Grade 0] or mild [Grade 1]) was achieved at 10, 15, 30, 45, 60, 90, and 120 minutes after the initial dose for all attacks.
Time Frame: Baseline and 10, 15, 30, 45, 60, 90, and 120 minutes post-dose (up to 24 weeks)
Population: FAS. The LOCF imputation method was used in this analysis.
Measure: Number; unit: percentage of attacks
Units Other Than Participants: number of moderate or severe attacks
Arm/Group | 20 mg Sumatriptan Nasal Powder | 100 mg Sumatriptan Tablet
Number analyzed (Participants) | 185 | 185
Number analyzed (number of moderate or severe attacks) | 509 | 532
percentage of attacks
  10 minutes post-dose | 13.8 | 11.5
  15 minutes post-dose | 27.9 | 20.9
  30 minutes post-dose | 53.8 | 38.7
  45 minutes post-dose | 65.0 | 53.9
  60 minutes post-dose | 72.1 | 62.6
  90 minutes post-dose | 77.4 | 72.0
  120 minutes post-dose | 79.6 | 76.9
Statistical Analysis 1: Comparison: 20 mg Sumatriptan Nasal Powder vs 100 mg Sumatriptan Tablet; Test type: Superiority or Other; p = 0.2426, ANCOVA; Odds Ratio (OR) = 1.24, 95% CI 2-sided [0.87 to 1.77] — 10 minutes post-dose
Statistical Analysis 2: Comparison: 20 mg Sumatriptan Nasal Powder vs 100 mg Sumatriptan Tablet; Test type: Superiority or Other; p = 0.0069, ANCOVA; Odds Ratio (OR) = 1.49, 95% CI 2-sided [1.12 to 1.99] — 15 minutes post-dose
Statistical Analysis 3: Comparison: 20 mg Sumatriptan Nasal Powder vs 100 mg Sumatriptan Tablet; Test type: Superiority or Other; p < 0.0001, ANCOVA; Odds Ratio (OR) = 1.94, 95% CI 2-sided [1.47 to 2.56] — 30 minutes post-dose
Statistical Analysis 4: Comparison: 20 mg Sumatriptan Nasal Powder vs 100 mg Sumatriptan Tablet; Test type: Superiority or Other; p = 0.0004, ANCOVA; Odds Ratio (OR) = 1.68, 95% CI 2-sided [1.26 to 2.23] — 45 minutes post-dose
Statistical Analysis 5: Comparison: 20 mg Sumatriptan Nasal Powder vs 100 mg Sumatriptan Tablet; Test type: Superiority or Other; p = 0.0008, ANCOVA; Odds Ratio (OR) = 1.60, 95% CI 2-sided [1.22 to 2.11] — 60 minutes post-dose
Statistical Analysis 6: Comparison: 20 mg Sumatriptan Nasal Powder vs 100 mg Sumatriptan Tablet; Test type: Superiority or Other; p = 0.0272, ANCOVA; Odds Ratio (OR) = 1.38, 95% CI 2-sided [1.04 to 1.83] — 90 minutes post-dose
Statistical Analysis 7: Comparison: 20 mg Sumatriptan Nasal Powder vs 100 mg Sumatriptan Tablet; Test type: Superiority or Other; p = 0.2085, ANCOVA; Odds Ratio (OR) = 1.21, 95% CI 2-sided [0.90 to 1.62] — 120 minutes post-dose

6. Secondary Outcome: Median Time to Pain Freedom
Description: Pain freedom is defined as a pain level reduced to none (Grade 0).
Time Frame: 120 minutes post-dose (up to 24 weeks)
Population: FAS. If the participant did not report pain freedom within 120 minutes post-dose, he/she was considered to be censored at the last non-missing result prior to the 120-minute time point.
Measure: Median (95% Confidence Interval); unit: minutes
Arm/Group | 20 mg Sumatriptan Nasal Powder | 100 mg Sumatriptan Tablet
Number analyzed (Participants) | 185 | 185
minutes | 91 [NA to NA] — The confidence interval is un-estimable due to the number of participants who were observed pain free at the post-dose time points. | 121 [91 to 121]

7. Secondary Outcome: Mean Change in Headache Severity From Baseline to 10, 15, 30, 45, 60, 90, and 120 Minutes Post-dose
Description: Participants were required to record their headache severity score in their e-diaries immediately before intake of study medication (Baseline) and at 10, 15, 30, 45, 60, 90, and 120 minutes post-dose. Participants graded their headaches on the following severity scale: 0, none; 1, mild; 2, moderate; 3, severe. Mean change from Baseline was calculated as the post-Baseline value minus the Baseline value.
Time Frame: Baseline and 10, 15, 30, 45, 60, 90, and 120 minutes post-dose (up to 24 weeks)
Population: FAS. The LOCF imputation method was used for this analysis. Results are from an ANCOVA model with treatment, period, and treatment sequence as fixed effects and participant as a random effect.
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | 20 mg Sumatriptan Nasal Powder | 100 mg Sumatriptan Tablet
Number analyzed (Participants) | 185 | 185
scores on a scale
  10 minutes post-dose | -0.11 (0.018) | -0.09 (0.018)
  15 minutes post-dose | -0.26 (0.029) | -0.18 (0.029)
  30 minutes post-dose | -0.56 (0.042) | -0.38 (0.042)
  45 minutes post-dose | -0.77 (0.049) | -0.60 (0.049)
  60 minutes post-dose | -0.93 (0.051) | -0.79 (0.051)
  90 minutes post-dose | -1.09 (0.052) | -0.98 (0.052)
  120 minutes post-dose | -1.19 (0.053) | -1.15 (0.053)
Statistical Analysis 1: Comparison: 20 mg Sumatriptan Nasal Powder vs 100 mg Sumatriptan Tablet; Test type: Superiority or Other; p = 0.3562, ANCOVA; Mean Difference (Final Values) = -0.02, 95% CI 2-sided [-0.06 to 0.02], Standard Error of Mean 0.021 — 10 minutes post-dose
Statistical Analysis 2: Comparison: 20 mg Sumatriptan Nasal Powder vs 100 mg Sumatriptan Tablet; Test type: Superiority or Other; p = 0.0063, ANCOVA; Mean Difference (Final Values) = -0.08, 94% CI 2-sided [-0.14 to -0.02], Standard Error of Mean 0.029 — 15 minutes post-dose
Statistical Analysis 3: Comparison: 20 mg Sumatriptan Nasal Powder vs 100 mg Sumatriptan Tablet; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = -0.19, 95% CI 2-sided [-0.26 to -0.11], Standard Error of Mean 0.039 — 30 minutes post-dose
Statistical Analysis 4: Comparison: 20 mg Sumatriptan Nasal Powder vs 100 mg Sumatriptan Tablet; Test type: Superiority or Other; p = 0.0005, ANCOVA; Mean Difference (Final Values) = -0.17, 95% CI 2-sided [-0.26 to -0.07], Standard Error of Mean 0.046 — 45 minutes post-dose
Statistical Analysis 5: Comparison: 20 mg Sumatriptan Nasal Powder vs 100 mg Sumatriptan Tablet; Test type: Superiority or Other; p = 0.0040, ANCOVA; Mean Difference (Final Values) = -0.14, 95% CI 2-sided [-0.24 to -0.05], Standard Error of Mean 0.048 — 60 minutes post-dose
Statistical Analysis 6: Comparison: 20 mg Sumatriptan Nasal Powder vs 100 mg Sumatriptan Tablet; Test type: Superiority or Other; p = 0.0333, ANCOVA; Mean Difference (Final Values) = -0.11, 95% CI 2-sided [-0.21 to -0.01], Standard Error of Mean 0.052 — 90 minutes post-dose
Statistical Analysis 7: Comparison: 20 mg Sumatriptan Nasal Powder vs 100 mg Sumatriptan Tablet; Test type: Superiority or Other; p = 0.4031, ANCOVA; Mean Difference (Final Values) = -0.04, 95% CI 2-sided [-0.15 to 0.06], Standard Error of Mean 0.052 — 120 minutes post-dose

8. Secondary Outcome: Mean Change From Baseline in Clinical Disability Score at 10, 15, 30, 45, 60, 90, and 120 Minutes Post-dose
Description: Participants were required to record their clinical disability score in their e-diaries immediately before intake of study medication (Baseline) and at 10, 15, 30, 45, 60, 90, and 120 minutes post-dose. Participants graded their disability on the following scale: 0, no disability, able to function normally; 1, performance of daily activities mildly impaired, can still do everything but with difficulty; 2, performance of daily activities moderately impaired, unable to do some things; 3, performance of daily activities severely impaired, cannot do all or most things, bed rest may be necessary. Mean change from Baseline was calculated as the post-Baseline value minus the Baseline value.
Time Frame: Baseline and 10, 15, 30, 45, 60, 90, and 120 minutes post-dose (up to 24 weeks)
Population: as for outcome 7
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | 20 mg Sumatriptan Nasal Powder | 100 mg Sumatriptan Tablet
Number analyzed (Participants) | 185 | 185
scores on a scale
  10 minutes post-dose | -0.08 (0.017) | -0.03 (0.017)
  15 minutes post-dose | -0.18 (0.025) | -0.09 (0.025)
  30 minutes post-dose | -0.42 (0.038) | -0.26 (0.038)
  45 minutes post-dose | -0.60 (0.046) | -0.43 (0.046)
  60 minutes post-dose | -0.73 (0.049) | -0.56 (0.049)
  90 minutes post-dose | -0.83 (0.052) | -0.72 (0.052)
  120 minutes post-dose | -0.92 (0.054) | -0.85 (0.054)
Statistical Analysis 1: Comparison: 20 mg Sumatriptan Nasal Powder vs 100 mg Sumatriptan Tablet; Test type: Superiority or Other; p = 0.0181, ANCOVA; Mean Difference (Final Values) = -0.04, 95% CI 2-sided [-0.08 to -0.01], Standard Error of Mean 0.019 — 10 minutes post-dose
Statistical Analysis 2: Comparison: 20 mg Sumatriptan Nasal Powder vs 100 mg Sumatriptan Tablet; Test type: Superiority or Other; p = 0.0003, ANCOVA; Mean Difference (Final Values) = -0.09, 95% CI 2-sided [-0.14 to -0.04], Standard Error of Mean 0.026 — 15 minutes post-dose
Statistical Analysis 3: Comparison: 20 mg Sumatriptan Nasal Powder vs 100 mg Sumatriptan Tablet; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = -0.16, 95% CI 2-sided [-0.23 to -0.09], Standard Error of Mean 0.035 — 30 minutes post-dose
Statistical Analysis 4: Comparison: 20 mg Sumatriptan Nasal Powder vs 100 mg Sumatriptan Tablet; Test type: Superiority or Other; p = 0.0001, ANCOVA; Mean Difference (Final Values) = -0.17, 95% CI 2-sided [-0.25 to -0.08], Standard Error of Mean 0.043 — 45 minutes post-dose
Statistical Analysis 5: Comparison: 20 mg Sumatriptan Nasal Powder vs 100 mg Sumatriptan Tablet; Test type: Superiority or Other; p = 0.0006, ANCOVA; Mean Difference (Final Values) = -0.16, 95% CI 2-sided [-0.26 to -0.07], Standard Error of Mean 0.047 — 60 minutes post-dose
Statistical Analysis 6: Comparison: 20 mg Sumatriptan Nasal Powder vs 100 mg Sumatriptan Tablet; Test type: Superiority or Other; p = 0.0189, ANCOVA; Mean Difference (Final Values) = -0.11, 95% CI 2-sided [-0.21 to -0.02], Standard Error of Mean 0.048 — 90 minutes post-dose
Statistical Analysis 7: Comparison: 20 mg Sumatriptan Nasal Powder vs 100 mg Sumatriptan Tablet; Test type: Superiority or Other; p = 0.1704, ANCOVA; Mean Difference (Final Values) = -0.07, 95% CI 2-sided [-0.17 to 0.03], Standard Error of Mean 0.050 — 120 minutes post-dose

9. Secondary Outcome: Number of Participants With Any Treatment-emergent Non-serious and Serious Adverse Event
Description: An adverse event is defined as any untoward medical occurrence associated with the use of an investigational product in humans, whether or not it is considered related to the investigational product. This includes any occurrence that was new in onset or aggravated in severity or frequency from the Baseline condition.
Time Frame: Baseline compared to Vist 2, 3 and 4
Population: Safety Analysis Set: all randomized participants who received at least 1 dose of either 20 mg sumatriptan nasal powder or 100 mg sumatriptan tablet
Measure: Number; unit: participants
Arm/Group | 20 mg Sumatriptan Nasal Powder | 100 mg Sumatriptan Tablet
Number analyzed (Participants) | 219 | 228
participants
  Treatment-emergent Adverse Event | 118 | 73
  Treatment-emergent Serious Adverse Event | 0 | 0

10. Secondary Outcome: Change From Baseline in Hemoglobin at Visit 3 (up to 12 Weeks) and Visit 4 (up to 24 Weeks)
Description: Change from Baseline in hemoglobin was assessed at Visit 3 (the start of Treatment Period 2) and Visit 4 (the end-of-study visit). Change from Baseline was calculated as the post-Baseline value minus the Baseline value. The Baseline value is the last non-missing value prior to or on the start date of Treatment Period 1.
Time Frame: Baseline and Visits 3 (up to 12 weeks) and 4 (up to 24 weeks)
Population: Safety Analysis Set. Only those participants with data available at Visit 3 and Visit 4 were assessed at that respective visit (indicated by n=X, X in the category titles).
Measure: Mean (Standard Deviation); unit: grams per Liter (g/L)
Groups:
- 20 mg Sumatriptan+PBO (TP1)/100 mg Sumatriptan+PBO (TP2): In Treatment Period 1 (<=12 weeks), participants received 20 milligrams (mg) sumatriptan nasal powder delivered intranasally with a bi-directional device and a placebo (PBO) tablet taken orally. After completing Treatment Period 1 (upon reaching 12 weeks or treating the fifth qualifying migraine headache in the treatment period, whichever came first), participants entered Treatment Period 2 (<=12 weeks), during which they received a 100 mg sumatriptan tablet taken orally and placebo (lactose) as a nasal powder administered into the nostril on the side of the migraine, followed by another administration into the other nostril. Participants were to treat <=5 qualifying migraine headaches during Treatment Period 2.
Arm/Group | 20 mg Sumatriptan+PBO (TP1)/100 mg Sumatriptan+PBO (TP2) | 100 mg Sumatriptan+PBO (TP1)/20 mg Sumatriptan+PBO (TP2)
Number analyzed (Participants) | 124 | 110
grams per Liter (g/L)
  Visit 3: number analyzed (Participants) | 109 | 95
  Visit 3 | -1.3 (6.07) | -1.3 (6.66)
  Visit 4 | -2.7 (6.58) | -0.8 (6.63)

11. Secondary Outcome: Change From Baseline in Hematocrit at Visit 3 (up to 12 Weeks) and Visit 4 (up to 24 Weeks)
Description: Change from Baseline in hematocrit (proportion of total blood volume that is composed of red blood cells) was assessed at Visit 3 (the start of Treatment Period 2) and Visit 4 (the end-of-study visit). Change from Baseline was calculated as the post-Baseline value minus the Baseline value.The Baseline value is the last non-missing value prior to or on the start date of Treatment Period 1.
Time Frame: Baseline and Visits 3 (up to 12 weeks) and 4 (up to 24 weeks)
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: proportion
Arm/Group | 20 mg Sumatriptan+PBO (TP1)/100 mg Sumatriptan+PBO (TP2) | 100 mg Sumatriptan+PBO (TP1)/20 mg Sumatriptan+PBO (TP2)
Number analyzed (Participants) | 124 | 110
proportion
  Visit 3, n=108, 94 | -0.002 (0.0204) | -0.005 (0.0222)
  Visit 4, n=124, 110 | -0.005 (0.0222) | -0.002 (0.0198)

12. Secondary Outcome: Change From Baseline in Red Blood Cell Count at Visit 3 (up to Week 12) and Visit 4 (up to Week 24)
Description: Change from Baseline in red blood cell count was assessed at Visit 3 (the start of Treatment Period 2) and Visit 4 (the end-of-study visit). Change from Baseline was calculated as the post-Baseline value minus the Baseline value. The Baseline value is the last non-missing value prior to or on the start date of Treatment Period 1.
Time Frame: Baseline and Visits 3 (up to 12 weeks) and 4 (up to 24 weeks)
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: 10^12 cells per Liter
Arm/Group | 20 mg Sumatriptan+PBO (TP1)/100 mg Sumatriptan+PBO (TP2) | 100 mg Sumatriptan+PBO (TP1)/20 mg Sumatriptan+PBO (TP2)
Number analyzed (Participants) | 124 | 110
10^12 cells per Liter
  Visit 3, n=109, 95 | -0.02 (0.227) | -0.04 (0.280)
  Visit 4, n=124, 110 | -0.05 (0.228) | -0.02 (0.209)

13. Secondary Outcome: Change From Baseline in White Blood Cell Count, Basinophils, Monocytes, Neutrophils, Lymphocytes, Eosinophils, and Platelets at Visit 3 (up to Week 12) and Visit 4 (up to Week 24)
Description: Change from Baseline in white blood cell (WBC) count, basinophils, monocytes, neutrophils, lymphocytes, eosinophils, and platelets was assessed at Visit 3 (the start of Treatment Period 2) and Visit 4 (the end-of-study visit). Change from Baseline was calculated as the post-Baseline value minus the Baseline value. The Baseline value is the last non-missing value prior to or on the start date of Treatment Period 1.
Time Frame: Baseline and Visits 3 (up to 12 weeks) and 4 (up to 24 weeks)
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: 10^9 cells per Liter
Arm/Group | 20 mg Sumatriptan+PBO (TP1)/100 mg Sumatriptan+PBO (TP2) | 100 mg Sumatriptan+PBO (TP1)/20 mg Sumatriptan+PBO (TP2)
Number analyzed (Participants) | 124 | 110
10^9 cells per Liter
  WBC Count, Visit 3, n=109, 95 | -0.10 (1.398) | -0.19 (1.381)
  WBC Count, Visit 4, n=124, 110 | -0.05 (1.477) | -0.09 (1.464)
  Basophils, Visit 3, n=108, 95 | 0.000 (0.0301) | 0.000 (0.0297)
  Basophils, Visit 4, n=124, 110 | 0.000 (0.0283) | -0.001 (0.0235)
  Monocytes, Visit 3, n=108, 95 | -0.030 (0.1356) | -0.022 (0.1160)
  Monocytes, Visit 4, n=124, 110 | -0.014 (0.1504) | -0.026 (0.1281)
  Neutrophils, Visit 3, n=108, 95 | -0.052 (1.2553) | -0.134 (1.1600)
  Neutrophils, Visit 4, n=124, 110 | -0.059 (1.4270) | -0.057 (1.2885)
  Lymphocytes, Visit 3, n=108, 95 | -0.049 (0.4702) | -0.038 (0.3892)
  Lymphocytes, Visit 4, n=124, 110 | 0.012 (0.4252) | -0.020 (0.3925)
  Eosinophils, Visit 3, n=108, 95 | -0.001 (0.0766) | 0.006 (0.0493)
  Eosinophils, Visit 4, n=124, 110 | 0.012 (0.1068) | 0.013 (0.0824)
  Platelets, Visit 3, n=109, 93 | -1.9 (29.14) | -8.2 (46.92)
  Platelets, Visit 4, n=123, 110 | -4.0 (27.92) | -7.5 (43.40)

14. Secondary Outcome: Change From Baseline in Urea at Visit 3 (up to Week 12) and Visit 4 (up to Week 24)
Description: Change from Baseline in urea was assessed at Visit 3 (the start of Treatment Period 2) and Visit 4 (the end-of-study visit). Change from Baseline was calculated as the post-Baseline value minus the Baseline value. The Baseline value is the last non-missing value prior to or on the start date of Treatment Period 1.
Time Frame: Baseline and Visits 3 (up to 12 weeks) and 4 (up to 24 weeks)
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: millimoles per Liter (mmol/L)
Arm/Group | 20 mg Sumatriptan+PBO (TP1)/100 mg Sumatriptan+PBO (TP2) | 100 mg Sumatriptan+PBO (TP1)/20 mg Sumatriptan+PBO (TP2)
Number analyzed (Participants) | 123 | 110
millimoles per Liter (mmol/L)
  Visit 3, n=108, 94 | 0.070 (1.2118) | 0.079 (1.2227)
  Visit 4, n=123, 110 | 0.156 (1.2840) | 0.308 (1.3674)

15. Secondary Outcome: Change From Baseline in Creatinine at Visit 3 (up to Week 12) and Visit 4 (up to Week 24)
Description: Change from Baseline in creatinine was assessed at Visit 3 (the start of Treatment Period 2) and Visit 4 (the end-of-study visit). Change from Baseline was calculated as the post-Baseline value minus the Baseline value. The Baseline value is the last non-missing value prior to or on the start date of Treatment Period 1.
Time Frame: Baseline and Visits 3 (up to 12 weeks) and 4 (up to 24 weeks)
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: micromoles per Liter (µmol/L)
Arm/Group | 20 mg Sumatriptan+PBO (TP1)/100 mg Sumatriptan+PBO (TP2) | 100 mg Sumatriptan+PBO (TP1)/20 mg Sumatriptan+PBO (TP2)
Number analyzed (Participants) | 123 | 110
micromoles per Liter (µmol/L)
  Visit 3, n=108, 94 | -1.9 (10.73) | -0.7 (6.59)
  Visit 4, n=123, 110 | -1.3 (11.77) | -0.6 (8.24)

16. Secondary Outcome: Change From Baseline in Alkaline Phosphatase (ALP) and Alanine Aminotransferase (ALT) at Visit 3 (up to Week 12) and Visit 4 (up to Week 24)
Description: Change from Baseline in ALP and ALT was assessed at Visit 3 (the start of Treatment Period 2) and Visit 4 (the end-of-study visit). Change from Baseline was calculated as the post-Baseline value minus the Baseline value. The Baseline value is the last non-missing value prior to or on the start date of Treatment Period 1.
Time Frame: Baseline and Visits 3 (up to 12 weeks) and 4 (up to 24 weeks)
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: International Units per Liter (IU/L)
Arm/Group | 20 mg Sumatriptan+PBO (TP1)/100 mg Sumatriptan+PBO (TP2) | 100 mg Sumatriptan+PBO (TP1)/20 mg Sumatriptan+PBO (TP2)
Number analyzed (Participants) | 123 | 110
International Units per Liter (IU/L)
  ALP, Visit 3, n=108, 94 | -0.5 (8.92) | 0.0 (6.78)
  ALP, Visit 4, n=123, 110 | -1.7 (9.92) | -1.0 (9.45)
  ALT, Visit 3, n=108, 94 | 0.4 (7.08) | 0.0 (8.86)
  ALT, Visit 4, n=123, 110 | 0.4 (6.83) | -0.9 (7.16)

17. Secondary Outcome: Change From Baseline in Aspartate Aminotransferase (AST) and Gamma Glutamyl Transferase (GGT) at Visit 3 (up to Week 12) and Visit 4 (up to Week 24)
Description: Change from Baseline in AST and GGT was assessed at Visit 3 (the start of Treatment Period 2) and Visit 4 (the end-of-study visit). Change from Baseline was calculated as the post-Baseline value minus the Baseline value. The Baseline value is the last non-missing value prior to or on the start date of Treatment Period 1.
Time Frame: Baseline and Visits 3 (up to 12 weeks) and 4 (up to 24 weeks)
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: International Units per Liter (IU/L)
Arm/Group | 20 mg Sumatriptan+PBO (TP1)/100 mg Sumatriptan+PBO (TP2) | 100 mg Sumatriptan+PBO (TP1)/20 mg Sumatriptan+PBO (TP2)
Number analyzed (Participants) | 123 | 110
International Units per Liter (IU/L)
  AST, Visit 3, n=108, 92 | -0.2 (5.26) | 0.5 (14.39)
  AST, Visit 4, n=123, 110 | 0.6 (7.88) | -1.2 (5.84)
  GGT, Visit 3, n=108, 94 | 0.8 (10.09) | 0.0 (7.05)
  GGT, Visit 4, n=123, 110 | 0.4 (10.31) | -0.7 (7.35)

18. Secondary Outcome: Change From Baseline in Total Bilirubin at Visit 3 (up to Week 12) and Visit 4 (up to Week 24)
Description: Change from Baseline in total bilirubin was assessed at Visit 3 (the start of Treatment Period 2) and Visit 4 (the end-of-study visit). Change from Baseline was calculated as the post-Baseline value minus the Baseline value. The Baseline value is the last non-missing value prior to or on the start date of Treatment Period 1.
Time Frame: Baseline and Visits 3 (up to 12 weeks) and 4 (up to 24 weeks)
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: Units per Liter (U/L)
Arm/Group | 20 mg Sumatriptan+PBO (TP1)/100 mg Sumatriptan+PBO (TP2) | 100 mg Sumatriptan+PBO (TP1)/20 mg Sumatriptan+PBO (TP2)
Number analyzed (Participants) | 123 | 110
Units per Liter (U/L)
  Visit 3, n=108, 94 | 0.2 (4.26) | -0.2 (2.96)
  Visit 4, n=123, 110 | -0.6 (4.09) | 0.2 (4.01)

19. Secondary Outcome: Change From Baseline in Albumin and Total Protein at Visit 3 (up to Week 12) and Visit 4 (up to Week 24)
Description: Change from Baseline in albumin and total protein was assessed at Visit 3 (the start of Treatment Period 2) and Visit 4 (the end-of-study visit). Change from Baseline was calculated as the post-Baseline value minus the Baseline value. The Baseline value is the last non-missing value prior to or on the start date of Treatment Period 1.
Time Frame: Baseline and Visits 3 (up to 12 weeks) and 4 (up to 24 weeks)
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: grams per Liter (grams/L)
Arm/Group | 20 mg Sumatriptan+PBO (TP1)/100 mg Sumatriptan+PBO (TP2) | 100 mg Sumatriptan+PBO (TP1)/20 mg Sumatriptan+PBO (TP2)
Number analyzed (Participants) | 123 | 110
grams per Liter (grams/L)
  albumin, Visit 3, n=108, 94 | -0.8 (2.82) | -0.9 (2.84)
  albumin, Visit 4, n=123, 110 | -0.9 (2.98) | -0.5 (2.62)
  total protein, Visit 3, n=108, 94 | -1.0 (3.75) | -1.2 (3.61)
  total protein, Visit 4, n=122, 110 | -1.2 (4.20) | -1.0 (3.35)

20. Secondary Outcome: Change From Baseline in Sodium, Potassium, Chloride, Calcium, and Glucose at Visit 3 (up to Week 12) and Visit 4 (up to Week 24)
Description: Change from Baseline in sodium, potassium, chloride, calcium, and glucose was assessed at Visit 3 (the start of Treatment Period 2) and Visit 4 (the end-of-study visit). Change from Baseline was calculated as the post-Baseline value minus the Baseline value. The Baseline value is the last non-missing value prior to or on the start date of Treatment Period 1.
Time Frame: Baseline and Visits 3 (up to 12 weeks) and 4 (up to 24 weeks)
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: mmoles/L
Arm/Group | 20 mg Sumatriptan+PBO (TP1)/100 mg Sumatriptan+PBO (TP2) | 100 mg Sumatriptan+PBO (TP1)/20 mg Sumatriptan+PBO (TP2)
Number analyzed (Participants) | 123 | 110
mmoles/L
  sodium, Visit 3, n=108, 94 | -0.3 (2.62) | -0.5 (2.24)
  sodium, Visit 4, n=122, 110 | -0.3 (2.76) | -0.2 (2.25)
  potassium, Visit 3, n=108, 94 | -0.08 (0.440) | -0.04 (0.404)
  potassium, Visit 4, n=122, 110 | -0.10 (0.411) | -0.00 (0.406)
  chloride, Visit 3, n=108, 94 | -0.1 (2.95) | 0.0 (2.39)
  chloride, Visit 4, n=122, 110 | 0.2 (2.62) | 0.2 (2.51)
  calcium, Visit 3, n=108, 94 | -0.019 (0.1017) | -0.016 (0.1043)
  calcium, Visit 4, n=123, 110 | -0.011 (0.1058) | -0.006 (0.0886)
  glucose, Visit 3, n=108, 94 | 0.34 (1.316) | 0.05 (0.930)
  glucose, Visit 4, n=123, 110 | 0.20 (1.063) | 0.24 (1.135)

21. Secondary Outcome: Change From Baseline in Urinalysis Values by Dipstick Method at Visit 3 (up to Week 12) and Visit 4 (up to Week 24)
Description: Change from Baseline in urinalysis values was assessed at Visit 3 (the start of Treatment Period 2) and Visit 4 (the end-of-study visit). Change from Baseline was calculated as the post-Baseline value minus the Baseline value. The Baseline value is the last non-missing value prior to or on the start date of Treatment Period 1.
Time Frame: Baseline and Visits 3 (up to 12 weeks) and 4 (up to 24 weeks)
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: pH
Arm/Group | 20 mg Sumatriptan+PBO (TP1)/100 mg Sumatriptan+PBO (TP2) | 100 mg Sumatriptan+PBO (TP1)/20 mg Sumatriptan+PBO (TP2)
Number analyzed (Participants) | 124 | 109
pH
  Visit 3, n=108, 95 | -0.04 (0.603) | -0.03 (0.720)
  Visit 4, n=124, 109 | 0.01 (0.664) | -0.07 (0.658)

22. Secondary Outcome: Number of Participants With the Indicated Amounts of Protein, Glucose, Ketones, Blood, and White Blood Cells (WBCs) in Urine at Baseline, Visit 3 (up to Week 12), and Visit 4 (up to Week 24)
Description: The Baseline value is the last non-missing value prior to or on the start date of Treatment Period 1. Data are based on standard reads, with "1+," "2+," and "3+" indicating increasing amounts of metabolites in urine.
Time Frame: Baseline and Visits 3 (up to 12 weeks) and 4 (up to 24 weeks)
Population: Safety Analysis Set
Measure: Number; unit: participants
Arm/Group | 20 mg Sumatriptan+PBO (TP1)/100 mg Sumatriptan+PBO (TP2) | 100 mg Sumatriptan+PBO (TP1)/20 mg Sumatriptan+PBO (TP2)
Number analyzed (Participants) | 133 | 129
participants
  Protein, Baseline, negative | 112 | 105
  Protein, Baseline, trace | 16 | 19
  Protein, Baseline, 1+ | 5 | 3
  Protein, Baseline, 2+ | 0 | 2
  Protein, Visit 3, negative | 92 | 75
  Protein, Visit 3, trace | 11 | 15
  Protein, Visit 3, 1+ | 4 | 5
  Protein, Visit 3, 2+ | 1 | 0
  Protein, Visit 4, negative | 104 | 90
  Protein, Visit 4, trace | 17 | 12
  Protein, Visit 4, 1+ | 3 | 6
  Protein, Visit 4, 2+ | 0 | 1
  Glucose, Baseline, negative | 132 | 126
  Glucose, Baseline, trace | 1 | 2
  Glucose, Baseline, 3+ | 0 | 1
  Glucose, Visit 3, negative | 107 | 94
  Glucose, Visit 3, trace | 0 | 1
  Glucose, Visit 3, 3+ | 1 | 0
  Glucose, Visit 4, negative | 122 | 108
  Glucose, Visit 4, trace | 0 | 1
  Glucose, Visit 4, 1+ | 1 | 0
  Glucose, Visit 4, 3+ | 1 | 0
  Ketones, Baseline, negative | 124 | 121
  Ketones, Baseline, trace | 7 | 7
  Ketones, Baseline, 1+ | 0 | 1
  Ketones, Baseline, 2+ | 2 | 0
  Ketones, Visit 3, negative | 102 | 88
  Ketones, Visit 3, trace | 5 | 6
  Ketones, Visit 3, 1+ | 1 | 0
  Ketones, Visit 3, 2+ | 0 | 1
  Ketones, Visit 4, negative | 119 | 101
  Ketones, Visit 4, trace | 3 | 8
  Ketones, Visit 4, 1+ | 2 | 0
  Blood, Baseline, negative | 116 | 116
  Blood, Baseline, trace | 7 | 4
  Blood, Baseline, 1+ | 2 | 3
  Blood, Baseline, 2+ | 5 | 1
  Blood, Baseline, 3+ | 3 | 5
  Blood, Visit 3, negative | 94 | 78
  Blood, Visit 3, trace | 4 | 6
  Blood, Visit 3, 1+ | 5 | 4
  Blood, Visit 3, 2+ | 2 | 2
  Blood, Visit 3, 3+ | 3 | 5
  Blood, Visit 4, negative | 111 | 94
  Blood, Visit 4, trace | 3 | 6
  Blood, Visit 4, 1+ | 1 | 5
  Blood, Visit 4, 2+ | 4 | 3
  Blood, Visit 4, 3+ | 5 | 1
  WBCs, Baseline, negative | 99 | 101
  WBCs, Baseline, trace | 12 | 8
  WBCs, Baseline, 1+ | 12 | 11
  WBCs, Baseline, 2+ | 7 | 5
  WBCs, Baseline, 3+ | 3 | 4
  WBCs, Visit 3, negative | 90 | 75
  WBCs, Visit 3, trace | 8 | 7
  WBCs, Visit 3, 1+ | 4 | 4
  WBCs, Visit 3, 2+ | 5 | 6
  WBCs, Visit 3, 3+ | 1 | 3
  WBCs, Visit 4, negative | 105 | 85
  WBCs, Visit 4, trace | 5 | 7
  WBCs, Visit 4, 1+ | 4 | 5
  WBCs, Visit 4, 2+ | 8 | 8
  WBCs, Visit 4, 3+ | 2 | 4

23. Secondary Outcome: Change From Baseline in Systolic Blood Pressure (SBP) and Diastolic Blood Pressure (DBP) at Visit 3 (up to Week 12) and Visit 4 (up to Week 24)
Description: Change from Baseline in SBP and DBP was assessed at Visit 3 (the start of Treatment Period 2) and Visit 4 (the end-of-study visit). Change from Baseline was calculated as the post-Baseline value minus the Baseline value. The Baseline value is the last non-missing value prior to or on the start date of Treatment Period 1.
Time Frame: Baseline and Visits 3 (up to 12 weeks) and 4 (up to 24 weeks)
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: millimeters of mercury (mmHg)
Arm/Group | 20 mg Sumatriptan+PBO (TP1)/100 mg Sumatriptan+PBO (TP2) | 100 mg Sumatriptan+PBO (TP1)/20 mg Sumatriptan+PBO (TP2)
Number analyzed (Participants) | 124 | 111
millimeters of mercury (mmHg)
  SBP, Visit 3, n=110, 95 | 0.1 (11.58) | 1.5 (11.46)
  SBP, Visit 4, n=124, 111 | 1.6 (11.52) | 2.0 (11.94)
  DBP, Visit 3, n=110, 95 | -0.2 (7.17) | 1.0 (8.89)
  DBP, Visit 4, n=124, 111 | 0.2 (7.42) | -0.2 (7.90)

24. Secondary Outcome: Change From Baseline in Pulse at Visit 3 (up to Week 12) and Visit 4 (up to Week 24)
Description: Change from Baseline in pulse was assessed at Visit 3 (the start of Treatment Period 2) and Visit 4 (the end-of-study visit). Change from Baseline was calculated as the post-Baseline value minus the Baseline value. The Baseline value is the last non-missing value prior to or on the start date of Treatment Period 1.
Time Frame: Baseline and Visits 3 (up to 12 weeks) and 4 (up to 24 weeks)
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | 20 mg Sumatriptan+PBO (TP1)/100 mg Sumatriptan+PBO (TP2) | 100 mg Sumatriptan+PBO (TP1)/20 mg Sumatriptan+PBO (TP2)
Number analyzed (Participants) | 124 | 111
beats per minute
  Visit 3, n=110, 95 | 0.1 (8.63) | 0.1 (9.24)
  Visit 4, n=124, 111 | -2.2 (9.07) | -0.2 (10.96)

25. Secondary Outcome: Number of Participants With the Indicated 12-lead Electrocardiogram (ECG) Findings at Baseline, Visit 3 (up to Week 12), and Visit 4 (up to Week 24)
Description: The Baseline value is the last non-missing value prior to or on the start date of Treatment Period 1. Clinical significance was determined by the Investigator (per clinical judgement). A categorization of "normal" or "abnormal" was made per the investigators' clinical judgment of the ECG, taking the participants' demographic characteristics and other medical conditions into account. CS = clinically significant. CNS = clinically not significant.
Time Frame: Baseline and Visits 3 (up to 12 weeks) and 4 (up to 24 weeks)
Population: Safety Analysis Set
Measure: Number; unit: participants
Arm/Group | 20 mg Sumatriptan+PBO (TP1)/100 mg Sumatriptan+PBO (TP2) | 100 mg Sumatriptan+PBO (TP1)/20 mg Sumatriptan+PBO (TP2)
Number analyzed (Participants) | 133 | 129
participants
  Baseline, normal; n=133, 129 | 96 | 99
  Baseline, abnormal, CS; n=133, 129 | 1 | 0
  Baseline, abnormal, CNS; n=133, 129 | 36 | 30
  Visit 3, normal; n=110, 95 | 79 | 70
  Visit 3, abnormal, CS; n=110, 95 | 0 | 0
  Visit 3, abnormal, CNS; n=110, 95 | 31 | 25
  Visit 4, normal; n=124, 111 | 90 | 73
  Visit 4, abnormal, CS; n=124, 111 | 0 | 1
  Visit 4, abnormal, CNS; n=123, 111 | 34 | 37

26. Secondary Outcome: Number of Participants With the Indicated Physical Examination Abnormalities at Baseline, Visit 3 (up to Week 12), and Visit 4 (up to Week 24)
Description: The Baseline value is the last non-missing value prior to or on the start date of Treatment Period 1. Clinical significance was determined by the Investigator (per clinical judgement). CS = clinically significant. CNS = clinically not significant.
Time Frame: Baseline and Visits 3 (up to 12 weeks) and 4 (up to 24 weeks)
Population: Safety Analysis Set
Measure: Number; unit: participants
Arm/Group | 20 mg Sumatriptan+PBO (TP1)/100 mg Sumatriptan+PBO (TP2) | 100 mg Sumatriptan+PBO (TP1)/20 mg Sumatriptan+PBO (TP2)
Number analyzed (Participants) | 133 | 129
participants
  Baseline, CS; n=133, 129 | 1 | 0
  Baseline, CNS; n=133, 129 | 132 | 129
  Visit 3, CS; n=110, 95 | 1 | 2
  Visit 3, CNS; n=110, 95 | 109 | 93
  Visit 4, CS; n=124, 111 | 0 | 0
  Visit 4, CNS; n=124, 111 | 124 | 111

27. Secondary Outcome: Number of Participants With the Indicated Concomitant Medications
Description: Concomitant medications are defined as non-study medications with a start or stop date between the first dose of study medication and the end of safety follow-up, inclusive. Derm. = dermatologic; incl. - including.
Time Frame: up to 24 weeks
Population: Safety Analysis Set
Measure: Number; unit: participants
Arm/Group | 20 mg Sumatriptan+PBO (TP1)/100 mg Sumatriptan+PBO (TP2) | 100 mg Sumatriptan+PBO (TP1)/20 mg Sumatriptan+PBO (TP2)
Number analyzed (Participants) | 219 | 228
participants
  Any concomitant medication | 218 | 226
  Agents acting on the renin-angiotensin system | 12 | 14
  Other therapeutic products | 2 | 2
  Allergens | 3 | 4
  Anabolic agents for systemic use | 1 | 1
  Analgesics | 143 | 148
  Anesthetics | 6 | 6
  Anti-acne preparations | 2 | 2
  Anti-Parkinson drugs | 3 | 3
  Antianemic preparations | 18 | 20
  Antibacterials for systemic use | 13 | 17
  Antibiotics and chemotherapeutics for derm. use | 0 | 2
  Antidiarrrheals, intestinal antiinflammatories | 7 | 6
  Antiemetics and antinauseants | 11 | 12
  Antiepileptics | 5 | 4
  Antigout preparations | 1 | 1
  Antihistamines for systemic use | 38 | 39
  Antiinflammatory and antirheumatic products | 135 | 143
  Antimyotics for systemic use | 1 | 3
  Antiobesity preparations, exluding diet products | 3 | 3
  Antiprotozoals | 0 | 1
  Antiseptics and disinfectants | 1 | 0
  Antithrombotic agents | 8 | 8
  Antivirals for systemic use | 2 | 3
  Beta blocking agents | 18 | 15
  Calcium channel blockers | 9 | 8
  Cardiac therapy | 1 | 1
  Corticosteroids for systemic use | 7 | 8
  Corticosteroids, dermatologic preparations | 1 | 1
  Cough and cold preparations | 8 | 9
  Diuretics | 6 | 7
  Drugs for acid related disorders | 22 | 23
  Drugs for functional gastrointestinal disorders | 5 | 3
  Drugs for obstructive airways diseases | 20 | 26
  Drugs for treatment of bone diseases | 1 | 1
  Drugs used in diabetes | 7 | 9
  Ectoparasiticides, incl. scabacides, insecticides | 1 | 0
  Gynecological antiinfectives and antiseptics | 1 | 2
  Immune sera and immunoglobulins | 1 | 1
  Laxatives | 4 | 3
  Lipid modifying agents | 23 | 20
  Mineral supplements | 20 | 22
  Muscle relaxants | 12 | 16
  Nasal preparations | 25 | 27
  Opthalmologicals | 7 | 6
  Other alimentary tract and metabolism products | 5 | 5
  Other dermatological preparations | 1 | 1
  Other gynecologicals | 21 | 21
  Other nervous system drugs | 3 | 3
  Otologicals | 1 | 0
  Psychoanaleptics | 57 | 60
  Psycholeptics | 31 | 31
  Sex hormones and modulators of the genital system | 62 | 59
  Thyroid therapy | 18 | 16
  Unspecified herbal and traditional medicine | 11 | 12
  Urologicals | 3 | 4
  Vaccines | 1 | 2
  Vitamins | 57 | 56

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events were collected from the first dose of investigational product through up to 24 weeks.
Description: Adverse events were collected in members of the Safety Analysis Set, comprised of all randomized participants who received at least 1 dose of either 20 mg sumatriptan nasal powder or 100 mg sumatriptan tablet.
Arm/Group | 20 mg Sumatriptan Nasal Powder | 100 mg Sumatriptan Tablet
Serious Adverse Events (participants affected / at risk) | 0/219 | 0/228
Other Adverse Events (participants affected / at risk) | 98/219 | 35/228
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 20 mg Sumatriptan Nasal Powder (N=219) | 100 mg Sumatriptan Tablet (N=228)
Nausea (Gastrointestinal disorders) | 9 | 7
Product taste abnormal (General disorders) | 57 | 9
Ear infection (Infections and infestations) | 1 | 3
Gastroenteritis viral (Infections and infestations) | 1 | 3
Sinusitis (Infections and infestations) | 3 | 4
Upper respiratory tract infection (Infections and infestations) | 9 | 8
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 3
Headache (Nervous system disorders) | 2 | 3
Nasal discomfort (Respiratory, thoracic and mediastinal disorders) | 34 | 3
Rhinalgia (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 4 | 0
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 6 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other